CLINICAL TRIAL: NCT06724679
Title: VRFR- Immersive Virtual Reality Use in a Spine Functional Restoration Program - A Feasibility Study
Acronym: VRFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Centre Hospitalier de l'Universite Laval (CHUL) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 49RC24_0176; 2024-A01741-46 (Other: ID-RCB - French-Health-Autorities)
Record Dates: First submitted 2024-11-29; First posted 2024-12-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low Back Pain
Keywords: Functionnal Restauration Program; Chronic low Back Pain; Immersive Virtual Reality

STUDY DESIGN:
Intervention Model Description: This study is a multicentric, prospective, exploratory interventional pilot trial aimed at assessing the feasibility of using an immersive VR device in a functional restoration program (FRP) for patients with chronic low back pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Utilisability of an immersive VR device in a functional restoration program (FRP) for patients with chronic low back pain.

INTERVENTIONS:
Other: Utilisability of an immersive VR device in a functional restoration program (FRP) for patients with chronic low back pain. — Patients participating will engage in three 20-minute VR sessions per week, in addition to the standard FRP program, for a duration of four to five weeks. The sessions will consist of a series of pre-programmed exercises designed to facilitate various trunk movements (flexion, extension, inclination, rotation) through exergames. Each exercise will last an average of 5 to 7 minutes. These exercises have been developed in collaboration between the company providing the VR device and the rehabilitation teams. Patients will be set up by a healthcare provider in a dedicated room for VR use. The provider will configure the device, assist the patient in donning it, and initiate the program, will remain present throughout the session to monitor for any adverse effect
  . While the specific exercises may vary, the total duration of the session will be 20 minutes, consisting of various exercises interspersed with breaks. The principal investigator will propose a standardized series of exercises,

SUMMARY:
This clinical trial investigates the feasibility of integrating immersive virtual reality (VR) technology into a functional restoration program (FRP) for patients with chronic low back pain (CLBP). The study aims to assess the acceptability, usability, and impact of a VR headset on both healthcare providers and patients participating in a group-based rehabilitation program. Chronic low back pain is a leading cause of functional disability worldwide and significantly impacts quality of life. Current rehabilitation strategies, including FRP, focus on improving physical functioning through multidisciplinary approaches. However, the role of emerging technologies, particularly VR, in enhancing these rehabilitation programs remains underexplored. VR has already shown promise in reducing chronic pain and improving motor abilities, but its application in a group rehabilitation context for CLBP is novel. The study will recruit healthcare providers and patients from several centers that are part of the Lombaction network. Participants will use a VR headset designed specifically to improve motor skills and reduce pain. The primary objective is to evaluate the acceptability of the VR device by healthcare providers and patients, as well as the usability and adherence to the VR program. Secondary objectives include assessing the impact of VR on kinesiophobia, pain, functional abilities, and motor imagery capabilities. This pilot study will provide valuable insights into the feasibility of incorporating VR into group-based rehabilitation programs, offering a foundation for larger comparative trials aimed at evaluating the long-term effectiveness of VR in improving rehabilitation outcomes for chronic low back pain.

DETAILED DESCRIPTION:
Study Overview: This multicentric, prospective, exploratory, interventional pilot study aims to assess the feasibility of integrating an immersive virtual reality (VR) headset into a functional restoration program (FRP) for patients with chronic low back pain (CLBP). Chronic low back pain is a leading cause of disability, and although current FRP approaches have demonstrated benefits, there is limited research on the integration of emerging technologies like VR into these rehabilitation programs. The primary focus of this study is to evaluate the acceptability and usability of VR technology among both healthcare providers and patients involved in group-based FRP rehabilitation. Secondary objectives include assessing the potential effects of VR on reducing kinesiophobia, improving motor imagery abilities, reducing pain, and enhancing overall functional capabilities. Study Objectives: Primary Objective: To assess the acceptability of the immersive VR headset for healthcare providers managing patients with CLBP in the context of a group-based FRP. Secondary Objectives: - To evaluate the usability and adherence of patients to the VR program.- To measure the effects of the VR sessions on kinesiophobia, motor imagery abilities, pain levels, and functional capacities. - To explore the factors influencing healthcare providers' and patients' acceptance of the VR device in this rehabilitation setting. Study Design: This study is designed as a pilot, multicentric, prospective, and interventional trial. Participants will be recruited from healthcare centers within the Lombaction network, a research-driven initiative for the management and evaluation of CLBP. Patients will receive standard FRP rehabilitation, along with 3 weekly VR sessions designed to enhance motor function and reduce pain through specific exercises targeting the spine and trunk. The VR system used is an immersive, wireless headset, designed to allow a wide variety of movement and requires no external controllers. Intervention: Patients will receive the standard FRP rehabilitation, which includes a combination of physiotherapy, hydrotherapy, occupational therapy, adapted physical activity, and therapeutic education workshops. The VR intervention will involve the use of a headset with pre-programmed exergames designed to improve trunk movement (flexion, extension, rotation, etc.). Each session will last 20 minutes, with exercises lasting 5-7 minutes each, aligned with current best practices in rehabilitation. The VR device is designed to be intuitive, requiring minimal setup, and will be used in a dedicated space at the rehabilitation center. In addition to the regular rehabilitation program, participants will engage in VR sessions three times per week for the duration of the FRP, which lasts 4-5 weeks. The VR sessions are intended to complement and enhance the physical rehabilitation by promoting movement, addressing kinesiophobia, and providing immersive, distraction-based pain management. Data Collection: Data will be collected at several points throughout the study: Baseline: At the beginning of the FRP, all patients will complete several questionnaires, including the Dallas Pain Questionnaire (DPQ), Tampa Scale for Kinesiophobia (TSK), Low Back Imagery Questionnaire, and a Visual Analog Scale (VAS) to assess pain. During the program: Patients will complete VAS assessments before and after each VR session. Weekly adherence data will be collected, noting whether the VR session was completed and the reasons for any missed sessions. End of the program: At the end of the FRP, participants will complete the same questionnaires as at baseline, as well as an additional acceptability questionnaire, and the System Usability Scale (SUS) to assess the usability of the VR device. Conclusion. This pilot study is designed to explore the feasibility of incorporating immersive VR technology into an existing FRP for patients with chronic low back pain. The results will provide valuable insights into the acceptability, usability, and potential therapeutic effects of VR in a group rehabilitation setting. If successful, this study could pave the way for larger trials to evaluate the long-term benefits of VR in the management of chronic low back pain and its integration into multidisciplinary rehabilitation programs.

ELIGIBILITY:
Caregiver Inclusion Criteria:

Caregivers involved in RFR programs at participating centers and likely to use the VR tool during the program.

Consent of the caregiver to participate in the study.

Patient Inclusion Criteria:

* Aged between 18 and 65 years.
* Diagnosed with chronic low back pain lasting more than three months, with secondary causes excluded.
* Candidates for integration into an RFR program at one of the participating centers.
* Affiliated with or beneficiaries of a social security scheme.
* Provide informed consent to participate in the study

Patient Exclusion Criteria:

* Presence of any other condition incompatible with the RFR program.
* Recent surgery or trauma (within the last month).
* Contraindications for using the VR device, including unstable epilepsy, facial trauma within the last three months, hearing or visual impairments, or previous experiences of pain, dizziness, or nausea triggered by VR device use.
* Visual impairments preventing the use of the VR device.
* Pregnancy or breastfeeding.
* Poor comprehension of the French language.
* Incarceration by judicial or administrative decision.
* Undergoing compulsory psychiatric treatment.
* Subject to legal protection measures.
* Incapable of providing informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
Acceptance of the VR system | 5 weeks (last day of Functional restoration program)
  a questionnaire based on the UTAUT 2 model

SECONDARY OUTCOMES:
Usability | 5 weeks (last day of Functional restoration program)
  System Usability Scale
Functional disability | day 1 and day 35 (First and Last day of the functional restauration program)
  Dallas Pain Questionnaire (DPQ)
Patient pain | day 1 and day 35 (First and Last day of the functional restauration program) and during VR session (before and after session)
  Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Romain CHAMPAGNE, MD, Principal Investigator — Hospital, Laval
Locations (5):
- France (5):
  - Les capucins, Angers
  - CH Cholet, Cholet
  - CH Laval, Laval
  - CHU Rennes, Rennes
  - Centre Hospitalier Bretagne Atlantique - Site de vannes, Vannes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Champagne R, Ali P, Ronzi Y, Dinomais M. Study protocol: use of virtual reality in a functional restoration programme for the spine-single-arm acceptance study. BMJ Open. 2025 Nov 26;15(11):e106366. doi: 10.1136/bmjopen-2025-106366. PMID 41298262